CLINICAL TRIAL: NCT01767766
Title: A Phase I Dose Escalation Study Evaluating the Safety and Efficacy of TGR 1202 in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: Evaluate the Safety and Efficacy of TGR 1202 in Patients With Relapsed or Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGR-1202-101 (HEMREF 31)
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Peripheral T-Cell Lymphoma; Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Peripheral; Hodgkin Disease | interventions — umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TGR-1202 (Experimental): TGR-1202 Daily Oral Dose
  Interventions: Drug: TGR-1202

INTERVENTIONS:
Drug: TGR-1202 — TGR-1202 Daily Oral Dose

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of TGR-1202 in patients with advanced hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Refractory to or relapsed after at least 1 prior treatment regimen;
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2;
* At least 18 years of age.

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days (limited palliative radiation is allowed ≥ 2 weeks);
* Autologous hematologic stem cell transplant within 3 months of study entry or Allogeneic hematologic stem cell transplant within 12 months;
* Known hepatitis B virus, hepatitis C virus or HIV infection;
* Previous therapy with GS-1101 (CAL-101), IPI-145 or any drug that specifically inhibits the PI3K or mTOR pathway;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose acceptable for participants | 28 days (1 cycle of therapy)
  To determine the incidence of adverse events, any potential abnormal laboratory results and any dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 1 year
  To assess the overall response rate (ORR) in patients with hematologic malignancies treated with TGR-1202

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, FACP, Study Chair — SCRI Development Innovations, LLC
Locations (7):
- United States (7):
  - TG Therapeutics Trial Site, Sarasota, Florida
  - TG Therapeutics Trial Site, Hackensack, New Jersey
  - TG Therapeutics Trial Site, New York, New York
  - TG Therapeutics Trial Site, Durham, North Carolina
  - TG Therapeutics Trial Site, Cincinnati, Ohio
  - TG Therapeutics Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Burris HA 3rd, Flinn IW, Patel MR, Fenske TS, Deng C, Brander DM, Gutierrez M, Essell JH, Kuhn JG, Miskin HP, Sportelli P, Weiss MS, Vakkalanka S, Savona MR, O'Connor OA. Umbralisib, a novel PI3Kdelta and casein kinase-1epsilon inhibitor, in relapsed or refractory chronic lymphocytic leukaemia and lymphoma: an open-label, phase 1, dose-escalation, first-in-human study. Lancet Oncol. 2018 Apr;19(4):486-496. doi: 10.1016/S1470-2045(18)30082-2. Epub 2018 Feb 20. PMID 29475723